CLINICAL TRIAL: NCT04872699
Title: Prevalence of COVID-19 in a French Dependent Care Facility for the Elderly and in a French Long-term Care Unit: Observational Study
Acronym: SPEED-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Sud Essonne (Other)
Responsible Party: Sponsor
Other Study IDs: SPEED-COVID19
Record Dates: First submitted 2021-05-02; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: elderly; COVID; SARS-COV-2; prevalence; dependant care; long-term unit
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serology testing, RT PCR — Periodic testings and testings with characteristic symptoms occur

SUMMARY:
The aim of this study is to evaluate the prevalence of COVID-19 among the residents and geriatric inpatients of the care facilities attached to the Centre Hospitalier Sud Essonne (a general hospital located in Ile-de-France, France), and the factors that are likely to influence this prevalence.

DETAILED DESCRIPTION:
Among people exposed to the COVID-19 (SARS-COV-2) pandemic, elderly people are considered as particularly vulnerable, especially those living in nursing homes or hospitalized. Furthermore, facilities / accommodations are registered among the main locations of COVID-19 clusters.

These observations have led the French government to establish specific protection measures and survey dependent care facilities for the elderly and long-term care units in the hospital.

With these new standards established, a long-term study of all the residents and geriatric inpatients of the care facilities attached to the Centre Hospitalier Sud Essonne (a general hospital located in Ile-de-France, France), can provide additional knowledge on COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* residents of the dependant care facility for the elderly
* inpatients of the long-term care unit
* from march, 2020 to december, 2021

Exclusion Criteria:

* opposition to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents and geriatric inpatients of the care facilities attached to the Centre Hospitalier Sud Essonne (a general hospital located in Ile-de-France, France), from march, 2020, to december, 2021, who are not opposed to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
General prevalence of COVID-19 | Through the study completion, an average of 12 months
  measures the prevalence of COVID-19 among the residents and geriatric inpatients, defined as resident and patients with positive serologic or RT-PCR test

SECONDARY OUTCOMES:
Number of asymptomatic residents/inpatients | Through study completion, an average of 12 months
  * no RT-PCR test or negative RT-PCR test and positive serologic test,
  * positive RT PCR and no symptoms.
Number of symptomatic residents/inpatients | Through study completion, an average of 12 months
  Positive RT-PCR test or serologic test with symptoms
Number of residents/inpatients with severe form of COVID-19 which led to an hospitalization | Through study completion, an average of 12 months
  Positive RT-PCR test or serologic test and hospitalization
Number of residents/inpatients infected with COVID-19 and hospitalized in a critical care unit | Through study completion, an average of 12 months
  Positive RT-PCR test or serologic test and hospitalization in critical care unit
Number of residents/inpatients infected with COVID-19 and deceased | Through study completion, an average of 12 months
  Positive RT-PCR test or serologic test and deceased
Number of residents/inpatients vaccinated against COVID-19 | Through study completion, an average of 12 months
  Positive RT-PCR test or serologic test and vaccinated with any authorized vaccine
Influencing factors of the prevalence of COVID-19 among residents/inpatients | Through study completion, an average of 12 months
  * age
  * sex
  * comorbidities
  * the context of the infection with COVID-19
  * vaccinated or not

CONTACTS AND LOCATIONS:
Overall Officials: Shidasp SIAMI, MD, PhD, Principal Investigator — Centre Hospitalier Sud Essonne
Locations (1):
- Centre Hospitalier Sud Essonne, Étampes, Essonne, France